CLINICAL TRIAL: NCT05840341
Title: Clinical Efficacy of QingyiHuaji Optimized Formula Combined With Standard Chemotherapy in the Treatment of Advanced Pancreatic Cancer: a Prospective, Multicenter, Randomized Controlled Clinical Study
Brief Title: Clinical Efficacy of QYHJ and Standard Chemotherapy in the Treatment of Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hao Chen, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2212267-7
Record Dates: First submitted 2023-04-09; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreatic Neoplasms; Traditional Chinese Medicine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): QingyiHuaji optimized formula combined with standard treatment
  Interventions: Drug: QingyiHuaji optimized formula
- Placebo group (Placebo Comparator): placebo combined with standard treatment
  Interventions: Drug: QingyiHuaji optimized formula

INTERVENTIONS:
Drug: QingyiHuaji optimized formula — Qingyihuaji Optimization Formula each bag contains: (1)Scutellaria barbata D. Don (Banzhilian); (2) Hedyotis diffusa Willd. (Sheshecao); (3) Amorphophallus rivieri Durieu (Sheliugu); (4) Amomi Fructus Rotundus (Doukou); (5) Gynostemma pentaphyllum (Thunb.) Makino (Jiaogulan); (6) Semen Coicis (Yiyiren); (7) Ganoderma lucidum (Curtis) P. Karst. (Lingzhi). One bag at a time, twice a day, rinsing with boiling water, continuous administration, oral administration in the morning and evening, every 3 weeks as a cycle.
  Other Names: standard chemotherapy

SUMMARY:
Our study is a prospective, multicenter, randomized controlled clinical study included patients with stage IV pancreatic ductal adenocarcinoma receiving gemcitabine-based first-line combination therapy according to the 2022 NCCN guidelines and with an estimated survival of > 3 months. According to reports and previous research results, we plan to include 306 subjects, and the subjects will divide into experimental group and the control group by a ratio of 1:1. All patients in the treatment group will receive QingyiHuaji optimized formula and standard treatment, and patients in the control group will receive placebo combined with standard treatment. Overall survival (OS) is defined as the primary endpoint, and progression-free survival (DFS), quality of life of cancer patients, and relief rate of TCM symptoms are considered as the secondary endpoint to observe the clinical efficacy of Qingyihuaji optimized formula combined with standard chemotherapy for stage IV pancreatic ductal adenocarcinoma. It will provide high-level evidence-based medical basis for the clinical effect of Qingyihuayi optimization prescription on pancreatic cancer with damp-heat accumulation syndrome. The hypothesis of this study is that the combination of Qingyihuaji optimized prescription with standard chemotherapy has the advantage of significantly prolonging the overall survival time, and is feasible and safe for the subjects diagnosed with stage IV pancreatic ductal adenocarcinoma by cytology or histology. The study lasted for 32 months, from 2023 April to December 2025.

DETAILED DESCRIPTION:
Pancreatic cancer is a digestive tract tumor with high malignancy and poor prognosis. The overall 5-year survival rate of early stage patients after surgery is less than 9%, while the median survival time of advanced stage patients is only 3-6 months. According to statistics, in 2020, there were about 420,000 new cases of pancreatic cancer worldwide, and about 410,000 deaths. In China, with the improvement of people's living standards and the progress of population aging, the incidence of pancreatic cancer is rising year by year, ranking 7th among men, and the mortality rate is 6th among men and 8th among women.

Due to its deep anatomical location, lack of typical clinical symptoms, and easy invasion and metastasis of tumors, pancreatic cancer is difficult to be detected in the early stage. More than 80% of patients are in local advanced stage or have distant metastasis at the time of diagnosis, thus losing the opportunity for radical surgery. Currently gemcitabine combined with albumin-binding paclitaxel regimen or FOLFIRINOX (fluorouracil, calcium leucovorin, irinotecan, oxaliplatin) regimen is the first-line chemotherapy regimen for pancreatic cancer.

However, pancreatic cancer has poor sensitivity to chemical and radiotherapy, and there has been little progress in targeted therapy and immunotherapy, resulting in no significant improvement in the survival rate of pancreatic cancer in recent decades. Meanwhile, the curative effect of other common tumors has made rapid progress. It is estimated by the NCI in the United States that if there is no breakthrough in the treatment of pancreatic cancer, pancreatic cancer will become the second largest tumor killer in human by 2030.

After nearly 20 years of dedicated research, the research team of Fudan University Shanghai cancer center, has carried out the integrated treatment mode of traditional Chinese and Western medicine to improve the survival of advanced pancreatic cancer patients, making the median OS of advanced pancreatic cancer patients reach the world leading level by 45% longer than that of chemotherapy alone, and the 3-year, 5-year survival rate reaches 15% and 6.2%, respectively. However, for patients with locally advanced unresectable pancreatic cancer without metastasis, how to improve their survival rate and quality of life is worth further researching.

The results suggest that QingyiHuayi formula has certain anti-tumor effect in advanced pancreatic cancer, and the combination of Qingyi Huayi formula with chemotherapy can prolong the survival period of patients, improve the clinical benefit rate, and may improve the therapeutic effective rate, without increasing the adverse reaction of radiotherapy and chemotherapy. The pathogenesis theory of cancer toxins puts forward that the pathogenesis of cancer toxins should be the core of syndrome differentiation, which solves the complicated and difficult problem of TCM tumor classification by disease differentiation. Four key points of clinical identification of cancer toxins pathogenesis were put forward to achieve the breakthrough of cancer virus identification and diagnosis technology bottleneck. To establish anti-cancer and detoxification treatment methods and classification of anti-cancer and detoxification Chinese medicines, and promote the clinical precision treatment and drug use of TCM tumors. Therefore, Qingyihuayi formula is a safe and effective treatment plan for advanced pancreatic cancer. After optimization, more clinical studies are needed to clarify the value of Qingyihuayi formula in the treatment of advanced pancreatic cancer and find more target groups of benefits.

In order to control random allocation and allocation hiding and ensure the science and standardization of randomized controlled trials, IWRS system of Beijing Biaoji Information Technology Co., Ltd. was used for randomization.

In order to ensure data multi-channel upload, safe storage, data desensitization and data sharing, as well as the accuracy of data entry and simple cleaning, the EDC system needs to be established. Beijing Biaozhi Information Technology Co., Ltd. is entrusted with the EDC system. It includes: ①EDC system; ②System supporting services: CRF annotation, eCRF establishment and testing, logic verification (logic verification plan, logic verification rule programming, logic verification rule testing), EDC training services; ③ Project management.

The median survival time of locally advanced pancreatic cancer is 4.43 months reported in relevant literatures, and the expected median survival time of the study group is 7.03 months. The test level (α) is set as 0.05, the test efficacy (1-β) as 0.80, and the expected shedding rate is 10%. After calculating by PASS software, a total of 306 patients are expected to be enrolled, and the experimental group and control group were randomly divided by 1:1, with 153 patients in the experimental group and 153 in the control group.

Descriptive statistical analysis will be used in this study. The measurement data are described by mean, standard deviation, median, lower quartile, upper quartile, minimum and maximum. Count data and rank data list frequency (component ratio) and rate. Describe the number of subjects enrolled in each group, and the number of cases dropped and eliminated. The final analysis of the study will be based on data collected by the subjects throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed Stage IV pancreatic ductal adenocarcinoma.
2. The expected survival time is >3 months;
3. Patients meet the standard treatment of gemcitabine - based first-line combination therapy recommended by the 2022 edition of the NCCN Pancreatic Cancer Guidelines;
4. Age above 18 years old and ≤75 years old;
5. ECOG physical state score 0-1;
6. Patients own adequate organ and bone marrow function, defined as neutrophils ≥1,500/ul, hemoglobin ≥ 8.0gm /dL, platelets ≥80,000/uL, serum creatinine < 2.0 mg/dL, bilirubin < 1.5 mg/dL, alanine aminotransferase < 3 times the upper limit of normal; If obstructive jaundice was allowed to enter the study after desicrin treatment, liver function markers were moderately relaxed to bilirubin < 2.5 mg/dL and alanine aminotransferase < 5 times the upper limit of normal.
7. Patients must have measurable lesions that meet the RECIST1.1 evaluation criteria. Bone scan abnormalities alone or osteolytic changes shown on plain radiographs cannot be measurable lesions, but can be evaluated in conjunction with bone scan abnormalities. Simple osteogenic bone metastases, pleural or peritoneal exudation, and radiation injury could not be considered as measurable lesions.
8. Patients who have not received "Qingyi Huayji Optimized formula " before (patients who have taken medicine for less than 2 weeks can be included at the discretion of the researchers) and who have received other traditional Chinese medicine treatment before must stop taking medicine 1 week before this study.
9. Female subjects of reproductive age must undergo a negative pregnancy test within 2 weeks prior to study drug initiation and be willing to use a medically approved highly effective contraceptive (e.g., intrauterine device, contraceptive or condom) during the study period and within 3 months after the last study drug administration; Male subjects with partners of women of reproductive age should agree to use effective contraceptive methods during the study period and within 3 months after the last study administration;
10. Patients is expected to possess good compliance, can understand and sign written informed consent, and willing to cooperate with the collection of TCM syndrome information;
11. SIRI value ≥0.8; SIRI = N × M/L, N, M, and L represent peripheral blood neutrophil, monocyte, and lymphocyte counts, respectively.

Exclusion Criteria:

1. Patients with ECOG score ≥2, who could not tolerate any antitumor therapy, or who could only receive the best supportive treatment were not considered for inclusion in this study.
2. The expected survival time < 3 months.
3. Other serious diseases or conditions, including deep vein thrombosis of the lower extremities, congestive heart failure (New York Heart Association Grade III or IV), unstable angina, etc.
4. Patients with co-infection requiring intravenous antibiotic treatment.
5. Pregnant or lactating women. Women of childbearing age who were unwilling or unable to use an acceptable method of contraception throughout the treatment period of this trial and within 12 weeks after the final administration of the study drug.
6. Known pancreatic neuroendocrine tumors, acinar cell carcinoma, intraductal papillary tumors and other types of pancreatic tumors.
7. Past or concurrent cancers with a primary focus or histologically distinct from pancreatic cancer, except cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Ta, Tis & T1). Any cancer that had been cured for more than 3 years prior to inclusion was admitted.
8. Those who are known to be allergic to components of Qingyihuaji optimized formula.
9. Unable to swallow Traditional Chinese medicine or untreated malabsorption syndrome, or unwilling to take Traditional Chinese medicine.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death from any cause, assess up to 24 months
  defined as the time from randomization to death from any cause. Subjects who are still alive at the time of final analysis or who have been lost to follow-up will be truncated at the last date of known survival.

SECONDARY OUTCOMES:
Disease Free Survival | From date of randomization until the date of first documented progression, assessed up to 24 months
  defined as the time from randomization to radiographic tumor progression or death from any cause. Subjects with no evidence of progress at the time of final analysis or who have been lost to follow-up will be truncated at the date of the last tumor evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chen, Study Director — Fudan University; Li Feng, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jun Qian, Study Chair — Affiliated Hospital of Nanjing University of Traditional Chinese Medicine; Aiguang Zhao, Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Affiliated Hospital of Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Sun D, Cao M, Li H, He S, Chen W. Cancer burden and trends in China: A review and comparison with Japan and South Korea. Chin J Cancer Res. 2020 Apr;32(2):129-139. doi: 10.21147/j.issn.1000-9604.2020.02.01. PMID 32410791
- [Background] Kamisawa T, Wood LD, Itoi T, Takaori K. Pancreatic cancer. Lancet. 2016 Jul 2;388(10039):73-85. doi: 10.1016/S0140-6736(16)00141-0. Epub 2016 Jan 30. PMID 26830752
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- [Background] Hua YQ, Wang P, Zhu XY, Shen YH, Wang K, Shi WD, Lin JH, Meng ZQ, Chen Z, Chen H. Radiofrequency ablation for hepatic oligometastatic pancreatic cancer: An analysis of safety and efficacy. Pancreatology. 2017 Nov-Dec;17(6):967-973. doi: 10.1016/j.pan.2017.08.072. Epub 2017 Sep 1. PMID 29129384
- [Background] Ouyang H, Wang P, Meng Z, Chen Z, Yu E, Jin H, Chang DZ, Liao Z, Cohen L, Liu L. Multimodality treatment of pancreatic cancer with liver metastases using chemotherapy, radiation therapy, and/or Chinese herbal medicine. Pancreas. 2011 Jan;40(1):120-5. doi: 10.1097/MPA.0b013e3181e6e398. PMID 20683216